CLINICAL TRIAL: NCT00943995
Title: TIW Growth Hormone Therapy in Children on Hemodialysis
Brief Title: Three Times Weekly (TIW) Growth Hormone Therapy in Children on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, John Mahan, Principal Investigator, Nationwide Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 907-M02R
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Failure, Chronic; Renal Dialysis
Keywords: End Stage Kidney Disease; Kidney Failure; Short stature; Growth Hormone therapy
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Dwarfism | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Other): Getting Growth Hormone therapy TIW instead of nightly in the Pediatric Tanner 1 Hemodialysis population.
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — 0.35 mg/Kg/week divided into 3 doses, each dose being given at the end of the dialysis treatment.
  Other Names: Nutropin AQ

SUMMARY:
Hypotheses:

1. The provision of thrice weekly subcutaneous (SQ) recombinant growth hormone (rGH) therapy to children receiving in-center hemodialysis (HD) will result in improved growth.
2. The provision of thrice weekly SQ rGH therapy to children receiving in-center HD will result in improved lean body mass, nutritional status and quality of life.

TIW rGH treatment regimen (0.35 mg/kg/week divided into 3 doses, each dose being given at the conclusion of the dialysis treatment) for up to 2 years; growth response, Dual energy X-ray absorptiometry (DEXA), and quality of life (QOL) will be measured. The goal is to enroll 20 children who are Tanner 1 with decreased height SDS and/or decreased height velocity standard deviation scoreS (SDS).

If this therapy is demonstrated to be efficacious and improves growth and QOL, this therapy could be easily implemented for all eligible children on HD, since parental acceptance should be better without having to administer the rGH at home and compliance for the child will be assured.

The investigators thus propose an important study that has the ability to advance their understanding and provide evidence for the best methods to promote growth in children on dialysis. The results of this study will result in important information that will be of value to the entire pediatric nephrologist community, including health care professionals, patients, and families. In a real sense, this study will build on the 2006 Consensus Conference guidelines for evaluation and treatment of growth failure in children with chronic kidney disease (CKD). This will provide evidence for critical management decisions that can help insure better growth opportunities to more children with CKD.

DETAILED DESCRIPTION:
Objectives/Aims:

1. To demonstrate the beneficial effects of thrice weekly SQ rGH Rx on growth in children on HD
2. To demonstrate the beneficial effects of thrice weekly SQ rGH Rx in terms of improved lean body mass, nutritional status and quality of life in children on HD

Study Design:

1. Study group - Provision of standard weekly dose of SQ rGH (0.35 mg/kg/week divided into 3 doses, each dose being given at the conclusion of dialysis therapy) for up to 2 years to growth retarded (Height SDS < -1.88 or Height velocity < -1.88 SD) children receiving HD who are naïve to rGH or who have not been on rGH for at least 12 months. Inclusion criteria are: medically cleared for SQ rGH Rx (14); growth potential based on Tanner stage 1 with open epiphyses on Bone Age radiographs (Bone age < 12 years); expected to require HD for at least 6 more months; at least 6 months of standardized historical pre-study anthropometric data (including stadiometer height). Exclusion criteria include all medical factors that indicate that rGH therapy should not be used (14), e.g., poor nutritional status, poorly controlled acidosis, poor dialysis adequacy (defined by Kt/V < 1.2), poorly controlled renal osteodystrophy (PTH > 800). Once the complicating factor is addressed and corrected, the child may be considered for the study.
2. SQ rGH to be provided in-center at the conclusion of dialysis session three times weekly for up to 24 months. SQ rGH dose to be adjusted based on dry (euvolemic) weight every month during the intervention.
3. Baseline and monitoring data obtained on each patient on SQ rGH Rx. This will include stadiometer measured height for at least 6 months prior to initiation of SQ rGH Rx to provide important baseline height and growth velocity to be used to determine magnitude of the response.
4. For children with suboptimal response after 6 months of standard SQ rGH Rx dose (annualized growth rate < 2 cm more than the preceding year), the rGH dose will be increased to 0.70 mg/kg/week divided into 3 doses (similar to the reported "pubertal" dosing regimen used in some GH deficient children).

Baseline data: Height (stadiometer), Weight, BMI, Height SDS, Height velocity SDS (historical past 6 months), Weight SDS, BMI SDS, Hb, BUN, nPCR, serum albumin, serum calcium, serum phosphorus, iPTH, electrolytes, high sensitivity CRP (as a marker of inflammation), dialysis adequacy (defined by single and double pool Kt/V - Kt/V is a unitless number used to quantify hemodialysis and peritoneal dialysis treatment adequacy: K - dialyzer clearance of urea, t - dialysis time, V - patient's total body water; in HD the target is 1.2), IGF-1, IGFBP-3, hip films and bone age (4,5,6,9). In addition, lean body mass/and fat mass will be assessed by DEXA (to standardize the determination of LBM, DEXA to be done mid week, after the dialysis treatment, to avoid the excess fluid commonly present after 2 days off dialysis each weekend) and quality of life will be assessed by the PedsQL 4.0 Generic Core Scales (10). The nutritional parameters that will be determined (wt/ht, ht SDS, BMI, nPCR and serum albumin) represent the currently used assessments of nutrition for these patients and have been validated as best measures of nutrition in children on dialysis (12).

Assessments to be repeated at the following intervals:

1. Height (stadiometer), Weight, Hgb, BUN, nPCR, serum albumin, serum calcium, phosphorus, and electrolytes, Kt/V - monthly
2. CRP, iPTH, IGF-1, IGFBP-3 - every 3 months
3. PedsQL - every 6 months
4. DEXA and Bone Age - yearly (and within 1 week of renal transplant if this occurs anytime 6 months after start of study) - DEXA and Bone Age results will be sent to Nationwide Children's and analyzed by our collaborating pediatric radiologist (Larry Binkovitz, MD).

ELIGIBILITY:
Inclusion Criteria:

* Chronic Renal Failure on Hemodialysis
* Tanner 1
* Bone Age <12
* Below the 3rd %tile for height or have growth velocity < 3rd %tile and are not on SQ rGH Rx
* At baseline, study population will also have to have documentation of normal thyroid status, secondary hyperparathyroidism will be controlled in acceptable range (iPTH < 800), adequate dialysis (Kt/V >1.2) and normal acid-base status.
* expected to be on hemodialysis at least 6 months

Exclusion Criteria:

* Anyone not meeting the inclusion criteria.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2010-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Primary Endpoints: Changes in Height SDS and Height velocity SDS | Will be monitored every 6 months

SECONDARY OUTCOMES:
Changes in Weight SDS, lean body mass, normalized protein catabolic rate and quality of life. | Will be monitored every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John D Mahan, MD, Principal Investigator — Nationwide Children's Hospital
Locations (5):
- United States (5):
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Children's Mercy Hospital, Kansas City, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - Children's Memorial Hermann Hospital-TMC, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Background] Feldt-Rasmussen B, Lange M, Sulowicz W, Gafter U, Lai KN, Wiedemann J, Christiansen JS, El Nahas M; APCD Study Group. Growth hormone treatment during hemodialysis in a randomized trial improves nutrition, quality of life, and cardiovascular risk. J Am Soc Nephrol. 2007 Jul;18(7):2161-71. doi: 10.1681/ASN.2006111207. Epub 2007 Jun 6. PMID 17554147
- [Background] Goldstein SL, Currier H, Watters L, Hempe JM, Sheth RD, Silverstein D. Acute and chronic inflammation in pediatric patients receiving hemodialysis. J Pediatr. 2003 Nov;143(5):653-7. doi: 10.1067/S0022-3476(03)00534-1. PMID 14615740
- [Background] Goldstein SL. Adequacy of dialysis in children: does small solute clearance really matter? Pediatr Nephrol. 2004 Jan;19(1):1-5. doi: 10.1007/s00467-003-1368-x. Epub 2003 Nov 22. PMID 14673636
- [Background] Goldstein SL, Brem A, Warady BA, Fivush B, Frankenfield D. Comparison of single-pool and equilibrated Kt/V values for pediatric hemodialysis prescription management: analysis from the Centers for Medicare & Medicaid Services Clinical Performance Measures Project. Pediatr Nephrol. 2006 Aug;21(8):1161-6. doi: 10.1007/s00467-006-0112-8. Epub 2006 May 17. PMID 16705459
- [Background] Gorman G, Frankenfield D, Fivush B, Neu A. Linear growth in pediatric hemodialysis patients. Pediatr Nephrol. 2008 Jan;23(1):123-7. doi: 10.1007/s00467-007-0631-y. Epub 2007 Oct 16. PMID 17934888
- [Background] Juarez-Congelosi M, Orellana P, Goldstein SL. Normalized protein catabolic rate versus serum albumin as a nutrition status marker in pediatric patients receiving hemodialysis. J Ren Nutr. 2007 Jul;17(4):269-74. doi: 10.1053/j.jrn.2007.04.002. PMID 17586426
- [Background] Kari JA, Rees L. Growth hormone for children with chronic renal failure and on dialysis. Pediatr Nephrol. 2005 May;20(5):618-21. doi: 10.1007/s00467-004-1801-9. Epub 2005 Mar 22. PMID 15782308
- [Background] Mahan JD, Warady BA; Consensus Committee. Assessment and treatment of short stature in pediatric patients with chronic kidney disease: a consensus statement. Pediatr Nephrol. 2006 Jul;21(7):917-30. doi: 10.1007/s00467-006-0020-y. Epub 2006 May 30. PMID 16773402
- [Background] Neu AM, Bedinger M, Fivush BA, Warady BA, Watkins SL, Friedman AL, Brem AS, Goldstein SL, Frankenfield DL. Growth in adolescent hemodialysis patients: data from the Centers for Medicare & Medicaid Services ESRD Clinical Performance Measures Project. Pediatr Nephrol. 2005 Aug;20(8):1156-60. doi: 10.1007/s00467-005-1889-6. Epub 2005 Jun 24. PMID 15977027